CLINICAL TRIAL: NCT00450658
Title: A Randomized, Double-Blind, Phase 3 Study of the Efficacy and Safety of HZT-501 in Subjects Requiring NSAID Treatment
Brief Title: Efficacy and Safety Study of HZT-501 in Reducing the Risk of Ibuprofen-associated Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HZ-CA-301
Record Dates: First submitted 2007-03-19; First posted 2007-03-22 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Peptic Ulcer
Keywords: ibuprofen; famotidine; ulcers; NSAIDS; pain; arthritis; chronic regional pain syndrome; chronic soft tissue pain; osteoarthritis; rheumatoid arthritis; chronic low back pain
MeSH Terms: conditions — Peptic Ulcer; Ulcer; Pain; Arthritis; Complex Regional Pain Syndromes; Osteoarthritis; Arthritis, Rheumatoid | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): HZT-501: Ibuprofen 800mg/Famotidine 26.6mg
  Interventions: Drug: HZT-501
- 2 (Active Comparator): Ibuprofen 800mg
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: HZT-501 — HZT-501: Ibuprofen 800mg/famotidine 26.6mg orally 3 times daily for 24 weeks
  Arms: 1
Drug: Ibuprofen — Ibuprofen 800mg orally 3 times daily for 24 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether HZT-501 is effective in reducing the rate of development of ibuprofen-associated ulcers in patients who require long-term daily use of ibuprofen.

DETAILED DESCRIPTION:
HZT-501 is a combination product including ibuprofen and the acid reducing agent famotidine. The study is designed to determine whether the combination product reduces the rate of ulcer development in subjects who require long-term daily use of ibuprofen.

Subjects will be assigned randomly, in approximately a 2:1 ratio, to treatment with either HZT-501 (ibuprofen 800 mg/famotidine 26.6 mg) or ibuprofen (800 mg) three times daily for a 24 week treatment period or until they develop either an endoscopically-diagnosed upper gastrointestinal ulcer and/or prohibitive toxicity. Subjects will visit the study center for Screening and at Weeks 4, 8, 16, and 24. Physical exams will be performed, and clinical laboratory measurements made, at selected times during the study. Endoscopic exams will be performed during Screening and at Weeks 8, 16, and 24. Subjects will be contacted four weeks following study completion.

Study with completed results acquired from Horizon in 2024

ELIGIBILITY:
Inclusion Criteria:

* Expected to require daily administration of a nonsteroidal anti-inflammatory drug (NSAID) for at least the coming six months for conditions such as osteoarthritis, rheumatoid arthritis, chronic low back pain, chronic regional pain syndrome, and chronic soft tissue pain.
* Did not use a NSAID within the 30 days prior to study entry

Exclusion Criteria:

* History of erosive esophagitis
* History of any of the following serious gastrointestinal complications:

  * perforation of ulcers,
  * gastric outlet obstruction due to ulcers,
  * gastrointestinal bleeding.
* Active cardiac, renal, and/or hepatic disease
* Current Helicobacter pylori (H. pylori) infection
* Use of an acid suppressant agent, misoprostol, or more than 325 mg/day of aspirin within the 14 days prior to study entry.
* Uncontrolled diabetes
* Uncontrolled hypertension
* Positive pregnancy test at screening
* Positive test at Screening for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Currently participating, or participation within 30 days prior to study entry, in an investigational drug study

Please note that there are other additional criteria. The study center will determine if patients meet all of the criteria.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Bello AE, Kent JD, Holt RJ. Gastroprotective efficacy and safety of single-tablet ibuprofen/famotidine vs ibuprofen in older persons. Phys Sportsmed. 2015 Jul;43(3):193-9. doi: 10.1080/00913847.2015.1066229. Epub 2015 Jul 13. PMID 26165391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center US study in which 80 sites recruited subjects between March 2007 and February 2008.
Pre-assignment Details: Following screening for eligibility and wash-out of restricted medications, subjects were assigned according to the treatment to which they were randomized in a 2:1 ratio (HZT-501:ibuprofen).
Groups:
- HZT-501: HZT-501: Ibuprofen 800mg/Famotidine 26.6mg tablets t.i.d.
- Ibuprofen: Ibuprofen 800mg tablets t.i.d.
Period: Overall Study
Arm/Group | HZT-501 | Ibuprofen
Started | 415 | 212
Completed | 272 | 122
Not Completed | 143 | 90
Not completed — Adverse Event | 24 | 15
Not completed — Withdrawal by Subject | 43 | 26
Not completed — Lost to Follow-up | 22 | 5
Not completed — UGI ulcer | 33 | 34
Not completed — misc | 21 | 10

BASELINE CHARACTERISTICS:
Groups:
- HZT-501: HZT-501: Ibuprofen 800mg/Famotidine 26.6mg
- Ibuprofen: Ibuprofen 800mg
- Total: Total of all reporting groups
Arm/Group | HZT-501 | Ibuprofen | Total
Number analyzed (Participants) | 415 | 212 | 627
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 342 | 173 | 515
  >=65 years | 73 | 39 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.0) | 55.7 (9.5) | 55.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 152 | 424
  Male | 143 | 60 | 203
Region of Enrollment [Number; unit: participants]
  United States | 415 | 212 | 627

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Develop Endoscopically-diagnosed Upper Gastrointestinal Ulcers Confirmed by Endoscopy.
Description: The primary efficacy endpoint was the number of subjects with upper gastrointestinal (i.e., gastric and/or duodenal) ulcer at any time throughout 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A subject is considered to have completed the study if all scheduled assessments up through the Week 24 visit have been performed.
Time Frame: 24 weeks
Population: All randomized subjects who received at least one dose of study drug and who underwent a baseline endoscopic examination and at least the Week 8 endoscopic examination.
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 380 | 190
participants | 40 [3.0 to 15.9] | 38 [3.0 to 15.9]
Statistical Analysis 1: Comparison: HZT-501 vs Ibuprofen; The primary efficacy endpoint was the proportion of subjects developing UGI (gastric and/or duodenal) ulcers throughout 24 weeks of treatment. A summary including cumulative frequency and percentage with associated 95% confidence intervals was produced for the observational incidences of UGI ulcers at 24 weeks. The cumulative proportion of subjects developing UGI ulcers at 24 weeks was analyzed using the CMH test stratified by use of low-dose aspirin and prior UGI ulcer history at randomization; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel; CMH test stratified by use of low-dose aspirin (Yes/No) and prior upper gastrointestinal ulcer history (Yes/No) at randomization; Risk Difference (RD) = 9.5, 95% CI 2-sided [3.0 to 15.9]

2. Secondary Outcome: Number of Subjects Who Develop Endoscopically-diagnosed Gastric Ulcers During the 24-week Treatment Period.
Description: The secondary efficacy endpoint was the number of subjects with gastric ulcer at any time throughout 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A subject is considered to have completed the study if all scheduled assessments up through the Week 24 visit have been performed.
Time Frame: 24 weeks
Population: The secondary efficacy endpoint was the number of subjects with gastric ulcer at any time throughout 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A subject is considered to have completed the study if all scheduled assessments up through the Week 24 visit were performed.
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 380 | 190
participants | 37 [1.9 to 14.4] | 34 [1.9 to 14.4]
Statistical Analysis 1: Comparison: HZT-501 vs Ibuprofen; Test type: Superiority or Other; p = 0.0051, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 8.2, 95% CI 2-sided [1.9 to 14.4]

3. Secondary Outcome: Number of Subjects Who Develop Endoscopically-diagnosed Duodenal Ulcers During the 24-week Treatment Period.
Description: The secondary efficacy endpoint was the number of subjects with duodenal ulcer at any time throughout the 24 weeks of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter with unequivocal depth. A subject is considered to have completed the study if all scheduled assessments up through the Week 24 visit have been performed.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 380 | 190
participants | 3 [0.8 to 7.1] | 9 [0.8 to 7.1]
Statistical Analysis 1: Comparison: HZT-501 vs Ibuprofen; The secondary efficacy endpoint was the proportion of subjects developing duodenal ulcers throughout 24 weeks of treatment. A summary including cumulative frequency and percentage with associated 95% confidence intervals was produced for the observational incidences of duodenal ulcers at 24 weeks. The cumulative proportion of subjects developing duodenal ulcers at 24 weeks was analyzed using the CMH test stratified by use of low-dose aspirin and prior UGI ulcer history at randomization; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel; CMH test stratified by use of low-dose aspirin and prior UGI ulcer history at randomization; Risk Difference (RD) = 3.9, 95% CI 2-sided [0.8 to 7.1]

4. Secondary Outcome: The Incidence Rate of NSAID-associated Serious Gastrointestinal Complications.
Description: The secondary efficacy endpoint was the number of subjects developing a NSAID-associated serious GI complication at any time throughout 6 months of treatment. A NSAID-associated serious GI complication was defined as a perforation of ulcers, gastric outlet obstruction due to ulcers, and/or GI bleeding.
Time Frame: 24 weeks
Population: All randomized subjects who received at least one dose of study drug and who underwent a baseline endoscopic exam. Subjects were assigned according to the treatment to which they received.
Measure: Number; unit: participants
Arm/Group | HZT-501 | Ibuprofen
Number analyzed (Participants) | 415 | 212
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Randomization through 24 weeks.
Description: Safety Population: All randomized subjects who received at least one dose of study drug and who underwent a baseline endoscopic examination. Subjects were assigned to the treatment to which they received; 2:1 randomization, HZT-501:ibuprofen.
Arm/Group | HZT-501 | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 11/415 | 4/212
Other Adverse Events (participants affected / at risk) | 220/415 | 116/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZT-501 (N=415) | Ibuprofen (N=212)
abscess (Infections and infestations) | 1 (1) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chest pain (General disorders) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
edema peripheral (General disorders) | 0 (0) | 1 (1)
esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
infection (Infections and infestations) | 1 (1) | 0 (0)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HZT-501 (N=415) | Ibuprofen (N=212)
abdominal distension (Gastrointestinal disorders) | 5 | 2
abdominal pain (Gastrointestinal disorders) | 7 | 4
abdominal pain upper (Gastrointestinal disorders) | 14 | 6
anemia (Blood and lymphatic system disorders) | 3 | 5
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 0
back pain (Musculoskeletal and connective tissue disorders) | 10 | 3
blood creatinine increased (Investigations) | 4 | 0
bronchitis (Infections and infestations) | 12 | 2
constipation (Gastrointestinal disorders) | 15 | 8
cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
depression (Psychiatric disorders) | 4 | 2
diarrhea (Gastrointestinal disorders) | 17 | 9
dyspepsia (Gastrointestinal disorders) | 17 | 18
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
edema peripheral (General disorders) | 6 | 3
flatulence (Gastrointestinal disorders) | 6 | 0
gastritis (Gastrointestinal disorders) | 7 | 3
gastroenteritis (Infections and infestations) | 4 | 0
gastroenteritis viral (Infections and infestations) | 2 | 3
gastroesophageal reflux (Gastrointestinal disorders) | 9 | 8
headache (Nervous system disorders) | 11 | 8
hypertension (Vascular disorders) | 11 | 4
influenza (Infections and infestations) | 8 | 1
influenza like illness (General disorders) | 4 | 0
insomnia (Psychiatric disorders) | 4 | 4
muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
nasopharyngitis (Infections and infestations) | 13 | 6
nausea (Gastrointestinal disorders) | 19 | 11
pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 2
rash (Skin and subcutaneous tissue disorders) | 3 | 3
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
sinusits (Infections and infestations) | 9 | 3
stomach discomfort (Gastrointestinal disorders) | 4 | 4
upper respiratory tract infection (Infections and infestations) | 16 | 11
urinary tract infection (Infections and infestations) | 3 | 3
vision blurred (Eye disorders) | 2 | 4
vomiting (Gastrointestinal disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI reserves the right to publish or otherwise make public the Study results provided that such communication occurs only after (i) the results of the multicenter Study in its entirety have been publicly disclosed by, or with consent of the sponsor or (ii) 18 months after conclusion of the Study at all sites, whichever comes first. Following this, PI can publish, present or use any non-confidential study results following Sponsor review. PI will not make public raw data or Case Reports.